CLINICAL TRIAL: NCT05584449
Title: Determining the Impact of a Curriculum for a Cancer Survivorship Group for Adolescents and Young Adults (AYA)
Brief Title: Group Curriculum for Improving Survivorship Outcomes in Adolescent and Young Adult Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-007844; NCI-2022-07825 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-10-11; First posted 2022-10-18 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (group curriculum) (Experimental): Participants attend an online group facilitated by two oncology social workers and receive information regarding coping with cancer survivorship as a young adult, as well as discuss survivorship issues/concerns with peers.
  Interventions: Other: Counseling; Procedure: Discussion; Other: Informational Intervention; Other: Medical Chart Review; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Counseling — Attend online group facilitated by two oncology social workers
  Other Names: Counseling Intervention
Procedure: Discussion — Discuss survivorship issues/concerns
  Other Names: Discuss
Other: Informational Intervention — Receive young adult cancer survivorship information
Other: Medical Chart Review — Ancillary studies
  Other Names: Chart Review
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies the effectiveness of a group curriculum in improving survivorship outcomes in adolescent and young adult (AYA) cancer survivors. Many AYA survivors typically do not feel prepared to re-enter "daily life" and would likely benefit from structured interventions to offer education and support in a timely manner as to prepare them for the challenges of life in survivorship. A 6-week group curriculum, designed to specifically meet the needs of AYA cancer survivors and facilitated by licensed social workers, may meet the unique needs of young adults who have survived a cancer diagnosis, and if so, the curriculum could be licensed and used across Mayo Clinic sites and potentially at other cancer centers nationwide.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Social workers will develop a curriculum to facilitate psychoeducational, skill-based, and process-oriented group for patients who have entered survivorship.

II. To determine if a specific 6 weeklong psychoeducational, skill-based, and process-oriented peer group curriculum results in improved quality of life for adolescents and young adult cancer survivors.

III. To demonstrate the feasibility of this curriculum to address the needs of this population.

OUTLINE:

Participants attend an online group facilitated by two oncology social workers and receive information regarding coping with cancer survivorship as a young adult, as well as discuss survivorship issues/concerns with peers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-39
* Is a patient of Mayo Clinic Arizona for oncologic care and/or follow-up
* History of cancer diagnosis
* Treated with curative intent
* Completed cancer treatment within 6 months to 2 years prior to group attendance
* Ability to read/write/speak English
* Ability to participate in a group setting
* Ability to commit to attending all six group meetings

Exclusion Criteria:

* Inability to read/write/speak English
* No internet or computer access
* Not receiving care at Mayo Clinic Arizona
* Currently receiving treatment for cancer
* Is unable to sit comfortably for 90 minutes
* Was not treated with curative intent
* Is on hospice care
* Co-morbid systemic illness or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessments

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2027-10-18 (Estimated); Study Completion 2027-10-18 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life | Baseline and 6 weeks
  Will be measured using the Quality of Life Patient/Cancer Survivor Version (QOL-CSV). The QOL-CSV is based on pre-existing versions of the City of Hope's QOL instrument. A pilot study conducted by Hassey-Dow and Farrell provided data which resulted in the revision of the QOL into 41 items that represent four domains of quality of life as pertaining to cancer survivorship: physical, psychological, social, and spiritual well-being. Only the psychological well-being, social concerns, and spiritual well-being components will be used. A two-sided paired t-test for the difference in the mean response will be conducted. A significance level of 0.05 will be used. If the data violate normality assumptions, a non-parametric alternative will be used. Additional summary statistics such as the proportion of participants who reported an improvement in QOL-CSV score may be used as appropriate.

SECONDARY OUTCOMES:
Change in well-being | Baseline and 6 weeks
  Will be measured using the Warwick-Edinburgh Mental Wellbeing scale (WEMWBS). 14 responses may be aggregated to provide a single score. The WEMWBS scale is a validated measurement of group mental well-being, which examines participants' hedonic and eudaemonic perspectives. A two-sided paired t-test for the difference in the mean response will be conducted. A significance level of 0.05 will be used. If the data violate normality assumptions, a non-parametric alternative will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Melody A Griffith, MSW, LISW, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials